CLINICAL TRIAL: NCT04894786
Title: Comparison of Mulligan Internal Rotation Mobilization and Post Isometric Relaxation Technique on Pain and Function in Athletes With Glenohumeral Internal Rotation Deficit
Brief Title: MIRM Versus PIRT in Athletes With Glenohumeral Internal Rotation Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/20/0108 Agha Salman Khan
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Glenohumeral Internal Rotation Deficit; Rotator Cuff Impingement; Internal Rotation Contracture-shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Internal Rotation Mobilization (Experimental): Mulligan Internal Rotation Mobilization & Sleeper Stretch
  Interventions: Other: Mulligan Internal Rotation Mobilization
- Post Isometric Relaxation Technique (Active Comparator): Post Isometric Relaxation Technique and Sleeper Stretch
  Interventions: Other: Post Isometric Relaxation Technique

INTERVENTIONS:
Other: Mulligan Internal Rotation Mobilization — Mulligan Internal Rotation Mobilization (MIRM) Sleeper Stretch The therapist places a web of his one hand around patient's axilla and thumb of another hand in the bent elbow and the glide will be applied to the head of the humerus down in the glenoid fossa using thumb while stabilizing the scapula with another hand. Therapist will ensures that the other hand is stabilizing up and inwards. While this distraction is taking place the patient internally rotated his shoulder with the help of another hand, at the same time his affected upper arm will abduct by therapist abdomen distracting the head of the humerus laterally. The hand in axilla acts as a fulcrum. Mulligan MWM will be applied for 3 days alternate days by following the rule of 3
  Arms: Mulligan Internal Rotation Mobilization
Other: Post Isometric Relaxation Technique — Post Isometric Relaxation Technique (PIRT) Sleeper Stretch The subject will be positioned supine on the treatment table with the shoulder and elbow, at 90 degree of abduction and flexion. The shoulder will be stabilized at the acromion process with one hand, and the other hand will be used to passively move the arm into internal rotation until the first barrier of motion will reached. The subject will be then instructed to perform a 5second isometric contraction of approximately 25% maximal effort in the direction of external rotation, against an opposing force provided at the distal forearm. Following the contraction, the subject will be instructed to internally rotate the arm toward the ground as a 30-second active assisted stretch will be applied. The subject will be instructed to relax, and a new movement barrier will then engage.
  Arms: Post Isometric Relaxation Technique

SUMMARY:
Glenohumeral internal rotation deficit (GIRD) is common physical deficiency found both teenager and overhead many sports for example baseball, cricket, and tennis. GIRD is generally categorized as simultaneous deficits of internal rotation (IR) and total arc of motion in the dominant side. GIRD causes increase muscle stiffness, capsular changes ( hyperplasia) , muscle imbalance leads to humeral retroversion. The objective of the study will be to Compare the effects of Mulligan internal rotation Mobilization and post isometric relaxation technique on Pain, Range of motion and function in athletes with Glenohumeral Internal Rotation Deficit

This study will be a Randomise Control trial and will be conducted Pakistan cricket board acedmy and in outpatient department of physical therapy, AL REHMAN Hospital Lahore . The study will be completed within the time duration of six months . Convenient sampling technique will be used to collect the data. A sample size of 14 patients will be taken in this study Comparison of Mulligan internal rotation Mobilization and post isometric relaxation technique on Pain and function in athletes with Glenohumeral Internal Rotation Deficit. Patients will be divided into two groups. (Group A will be treated with mulligan MWM AND Sleeper stretch whereas Group B will be treated with post isometic relaxtion technique and sleeper stretch ). SPADI score will be used to ask some questions related to patients symptoms and daily activities and Numeric pain rating scale will be used to measure pain intensity. UNIVERSAL GONIOMETER will be used to measure ROM of shoulder joint All participants of the study will fill the SPADI score and Numeric pain rating scale on day 1 as pre treatment values and at the end of week 2 as post treatment values respectively . The collected data will be analyzed on SPSS 25.

DETAILED DESCRIPTION:
Glenohumeral internal rotation deficit (GIRD) is common physical deficiency found both teenager and overhead many sports for example baseball, cricket, and tennis. GIRD is generally categorized as simultaneous deficits of internal rotation (IR) and total arc of motion in the dominant side.

Tight posterior glenohumeral capsule and posterior muscles such as the posterior deltoid, infraspinatus, and teres minor muscles can leads to GIRD although mechanism is not clear yet. Few research authors propose that repetitive tensile stress to posterior structures in the follow-through phase in throwing movements could lead to inflammation, scar formation, and following tightness in posterior tissues, resulting in PST and GIRD.

Tightness of the posterior shoulder may be a common factor in many shoulder conditions, including impingement syndrome, rotator cuff tears, and labral lesions.Posterior shoulder tightness may cause alterations in shoulder motion or muscle flexibility that are thought to increase risk of injury in athletes.

GIRD causes increase muscle stiffness, capsular changes ( hyperplasia ) , muscle imbalance leads to humeral retroversion.Due to the influence of tightness of the posterior glenohumeral soft tissues on glenohumeral and shoulder kinematics stretching of the posterior glenohumeral tissues to restore glenohumeral IR ROM is a common aspect of shoulder rehabilitation.

GIRD can be measured as the difference in the maximum humeral internal rotation angle between the dominant (throwing) and non-dominant (non-throwing) limbs. A difference of 10-17 degree of internal rotation is common in the dominant arm of throwing athletes who have not suffered any shoulder injury. GIRD greater than 25° has been associated with injuries such as superior labral lesions, subacromial impingement, and pathological internal impingement in the throwing shoulder in dictating a need for investigation of preventative and corrective interventions to restore GHJ internal rotation ROM.

Manual Physical thearpy approaches are very effective in treatment of many musculoskeletal issues. Mulligan manual techniques Introduced by Brain mulligan are very useful treating and correcting joint dysfunction. The mobilization with movement technique has its own parameter. It is done with both therapist patient participation i.e. passive glide is done by physiotherapist at peripheral joint meanwhile patient performs pain free physiologic movement. The stamp of mobilization with movement (MWM) technique is pain should be decreased after the application of technique.

Muscle energy techniques are basically soft tissue osteopathic manipulation which is performed precisely and in controlled manners, patient do isotonic or isometric contractions , they are very useful in function and reduce the pain . MET are mostly indicated in to decrease pain, stretch tight muscles and fascia, reduce muscle tonus, improve local circulation, strengthen weak musculature and mobilize joint restrictions . This leads to improved postural alignment and the restoration of proper joint biomechanics and functional movement.

As per as researcher's Knowledge most of the studies were conducted on over all mobility of shoulder, only few studies worked purely on internal rotation deficit. so this study will be benficient for GIRD.The rationale of this study will be to check the additive effects of Mulligan internal roation mobilization on Pain, Range of motion and function in athletes with Glenohumeral Internal Rotation Deficit beside the application of sleeper stretch a conventional protocol.

In 2018 Sreenivasu Kotagiri and his colleagues conduced a study on effectiveness of Mobilization with Exercise V/S Mulligan Internal Rotation MWM with Stretching in Patient with Glenohumeral Internal Rotation Deficit .They founded mulligan mobilization with posterior capsule stretching is more effective in improving range of motion and function when compared to mobilization with shoulder stabilization exercises alone.

In 2016 Sonakshi Sehgal and her colleague conducted a study to measure the effect muscle energy technique(MET) for the glenohumeral joint external rotators to improve the range of motion and strength of internal rotators in athletes with glenohumeral internal rotation deficit (GIRD). They found that MET can be used to treat limited glenohumeral internal rotation in athletes with GIRD. The study concluded that the treatment showed remarked improvement in the range of motion and strength of internal rotators in athletes with GIRD. Therefore the technique can be used in acute cases of posterior shoulder tightness to prevent the occurrence of other shoulder injuries.

In 2010 Robert C. Manske, and his colleagues worked on Comparison of Stretching Versus Stretching and Joint Mobilization for Posterior Shoulder Tightness Measured by Internal Rotation Motion Loss they concluded cross-body stretch and cross-body stretch plus joint mobilization ,both may be beneficial for those with limited internal rotation range of motion.

In 2013 Hafiz Sheraz Arshad and his colleagues worked on comparison of Mulligan Mobilization with Movement and End-Range Mobilization Following Maitland Techniques in Patients with Frozen Shoulder in Improving Range of Motion, they concluded that end range mobilization following maitland are equally effective as that of mobilization with movement exercises. Effectiveness of end range mobilization following maitland for increasing range of motion and improving pain. This supported their usefulness in improving quality of life due to shoulder dysfunction such as frozen shoulder.

As per as researcher's Knowledge most of the studies were conducted on over all mobility of shoulder, only few studies worked purely on internal rotation deficit. so this study will be benficient for GIRD.The rationale of this study will be to check the additive effects of Mulligan internal roation mobilization on Pain, Range of motion and function in athletes with Glenohumeral Internal Rotation Deficit beside the application of sleeper stretch a conventional protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects within the age group 18-35 years will be taken.
* Both male and female will be taken.
* Subjects with glenohumeral internal rotation deficit will be taken.
* Subjects with minimum 50% reduction in the internal rotation range of motion will be taken compared to the unaffected side.
* Subjects with shoulder abduction ROM at least 90 degrees
* Subjects with shoulder Extension ROM at least 20 degrees
* Subjects with positive lift-off test and belly compression test

Exclusion Criteria:

* History of shoulder surgery
* Any Shoulder joint complex fracture
* Frozen shoulder (Adhesive capsulitis)
* post traumatic and rotator cuff tear
* neurological deficit affecting shoulder
* Pain or disorder of cervical spine
* Osteoporosis, Malignancies ,Open wound and Pregnancy
* Rheumatoid arthritis
* a recent steroid injection and previous manipulation under anesthesia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE | 2 weeks
  NPRS is anchored by terms describing pain severity extremes. The 11 -point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable
Shoulder Pain and Disability Index (SPADI) | 2 weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
Universal Goniometer | 2 weeks
  Universal goniometer will be used to measure Shoulder internal rotation range of motion .

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Study Chair — Riphah International University
Locations (1):
- Al Rehman Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manske RC, Meschke M, Porter A, Smith B, Reiman M. A randomized controlled single-blinded comparison of stretching versus stretching and joint mobilization for posterior shoulder tightness measured by internal rotation motion loss. Sports Health. 2010 Mar;2(2):94-100. doi: 10.1177/1941738109347775. PMID 23015927
- [Background] Kotagiri N, Cooper ML, Rettig M, Egbulefu C, Prior J, Cui G, Karmakar P, Zhou M, Yang X, Sudlow G, Marsala L, Chanswangphuwana C, Lu L, Habimana-Griffin L, Shokeen M, Xu X, Weilbaecher K, Tomasson M, Lanza G, DiPersio JF, Achilefu S. Radionuclides transform chemotherapeutics into phototherapeutics for precise treatment of disseminated cancer. Nat Commun. 2018 Jan 18;9(1):275. doi: 10.1038/s41467-017-02758-9. PMID 29348537
- [Background] Sehgal R, Cheung CX, Hills T, Waris A, Healy D, Khan T. Perforated jejunal diverticulum: a rare case of acute abdomen. J Surg Case Rep. 2016 Oct 7;2016(10):rjw169. doi: 10.1093/jscr/rjw169. PMID 27765806
- [Background] Wilk KE, Macrina LC, Fleisig GS, Porterfield R, Simpson CD 2nd, Harker P, Paparesta N, Andrews JR. Correlation of glenohumeral internal rotation deficit and total rotational motion to shoulder injuries in professional baseball pitchers. Am J Sports Med. 2011 Feb;39(2):329-35. doi: 10.1177/0363546510384223. Epub 2010 Dec 4. PMID 21131681
- [Background] Tokish JM, Curtin MS, Kim YK, Hawkins RJ, Torry MR. Glenohumeral internal rotation deficit in the asymptomatic professional pitcher and its relationship to humeral retroversion. J Sports Sci Med. 2008 Mar 1;7(1):78-83. eCollection 2008. PMID 24150137
- [Background] Keller RA, De Giacomo AF, Neumann JA, Limpisvasti O, Tibone JE. Glenohumeral Internal Rotation Deficit and Risk of Upper Extremity Injury in Overhead Athletes: A Meta-Analysis and Systematic Review. Sports Health. 2018 Mar/Apr;10(2):125-132. doi: 10.1177/1941738118756577. Epub 2018 Jan 30. PMID 29381423